CLINICAL TRIAL: NCT00698581
Title: An International, Double-blind, Randomized, Multi-center, Parallel Group, Historical-control Conversion to Monotherapy Study to Evaluate the Efficacy and Safety of Brivaracetam in Subjects (≥ 16 to 75 Years Old) With Partial Onset Seizures With or Without Secondary Generalization
Brief Title: A Double-blind, Randomized Conversion to Monotherapy Study to Evaluate the Efficacy and Safety of Brivaracetam in Subjects (≥ 16 to 75 Years Old) With Partial Onset Seizures
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: An interim analysis revealed the study was unlikely to attain a positive outcome for the efficacy analysis. No safety concerns were detected.
Sponsor: UCB Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: N01276; 2008-000144-14 (EudraCT Number)
Expanded Access: NCT03532516 (Available)
Record Dates: First submitted 2008-06-12; First posted 2008-06-17 (Estimated); Results first posted 2016-04-13 (Estimated); Last update posted 2018-07-11 (Actual); Status verified 2018-03

CONDITIONS: Epilepsy
Keywords: Epilepsy; Monotherapy; Partial Onset Seizures; Adults and Adolescents
MeSH Terms: conditions — Epilepsy | interventions — brivaracetam

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Brivaracetam 50 mg (Experimental): 50 mg/day
  Interventions: Drug: Brivaracetam
- Brivaracetam 100 mg (Experimental): 100 mg/day
  Interventions: Drug: Brivaracetam

INTERVENTIONS:
Drug: Brivaracetam — 25 mg tablet - 50 mg daily for 17 weeks (or 21 weeks if down-titrated (50 mg > 20 mg) for subjects not participating in the follow-up study)
  Other Names: ucb 34714
  Arms: Brivaracetam 50 mg
Drug: Brivaracetam — 25 mg tablet - 100 mg daily for 17 weeks (or 21 weeks if down-titrated (100 mg > 50 mg > 20 mg) for subjects not participating in the follow-up study)
  Other Names: ucb 34714
  Arms: Brivaracetam 100 mg

SUMMARY:
Antiepileptic drugs (AEDs) are the main treatment for epilepsy; however, only a limited number of AEDs are approved for use as monotherapy. The objective of this study is to evaluate the efficacy of Brivaracetam (BRV) in the conversion of partial onset seizure patients from combination treatment to monotherapy

ELIGIBILITY:
Inclusion Criteria:

* Subjects from 16 to 75 years, both inclusive
* Well-characterized focal epilepsy or epileptic syndrome
* Subjects having at least 2 but not exceeding 40 partial onset seizures, whether or not secondarily generalized per 4 weeks during the 8-week Baseline Period
* Subjects on a stable dose of at least 1 but no more than 2 concomitant Antiepileptic Drugs (AEDs) with the second AED ≤ 50 % of the minimum recommended maintenance dose

Exclusion Criteria:

* Seizure type IA non-motor as only seizure type
* History or presence of seizures occurring too frequently or indistinctly separated to be reliably counted during the 6 months preceding Visit 1 or during Baseline
* Other serious uncontrolled disease

Ages: 16 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2008-08; Primary Completion 2010-01 (Actual); Study Completion 2010-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — +1 877 822 9493 (UCB)
Locations (53):
- United States (26):
  - Phoenix, Arizona
  - Fresno, California
  - Pasadena, California
  - Denver, Colorado
  - Miami, Florida
  - Orlando, Florida
  - Conyers, Georgia
  - Macon, Georgia
  - Peoria, Illinois
  - Lexington, Kentucky
  - Burlington, Massachusetts
  - Las Vegas, Nevada
  - Summit, New Jersey
  - Mineola, New York
  - New York, New York
  - The Bronx, New York
  - Hickory, North Carolina
  - Kettering, Ohio
  - Oklahoma City, Oklahoma
  - Germantown, Tennessee
  - Austin, Texas
  - Dallas, Texas
  - Houston, Texas
  - Danville, Virginia
  - Charleston, West Virginia
  - Waukesha, Wisconsin
- Australia (6):
  - Chatswood, New South Wales
  - Adelaide, South Australia
  - Clayton, Victoria
  - Fitzroy, Victoria
  - Parkville, Victoria
  - West Heidelberg, Victoria
- Belgium (2):
  - Ghent
  - Kortrijk
- Canada (5):
  - Calgary, Alberta
  - Edmonton, Alberta
  - Toronto, Ontario
  - Windsor, Ontario
  - Sakaskatoon, Saskatchewan
- Czechia (6):
  - Brno
  - Litomyšl
  - Ostava
  - Ostrava-Trebovice
  - Prague
  - Praha-4
- Germany (4):
  - Aschaffenburg
  - Halle
  - Mainz
  - Regensburg
- Sweden (4):
  - Gothenburg
  - Lund
  - Stockholm
  - Uppsala

REFERENCES:
- [Result] Arnold S, Badalamenti V, Diaz A, Gasalla T, McShea C, Whitesides J, Fakhoury T. Conversion to brivaracetam monotherapy for the treatment of patients with focal seizures: Two double-blind, randomized, multicenter, historical control, Phase III studies. Epilepsy Res. 2018 Mar;141:73-82. doi: 10.1016/j.eplepsyres.2018.02.005. Epub 2018 Feb 12. PMID 29486396

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study started to enroll patients in August 2008 and concluded in February 2010.
Pre-assignment Details: The Participant Flow refers to the Randomized Set (RS). Subjects withdrawn due to meeting an exit criterion are included in the count of early discontinuations with a reason of "Adverse Event" or "Lack of efficacy" as reported by the Investigator.
Groups:
- Brivaracetam 50 mg/Day: Brivaracetam: 25 mg tablet - 50 mg daily for 17 weeks (or 21 weeks if down-titrated (50 mg > 20 mg) for subjects not participating in the follow-up study)
- Brivaracetam 100 mg/Day: Brivaracetam: 25 mg tablet - 100 mg daily for 17 weeks (or 21 weeks if down-titrated (100 mg > 50 mg > 20 mg) for subjects not participating in the follow-up study)
Period: Overall Study
Arm/Group | Brivaracetam 50 mg/Day | Brivaracetam 100 mg/Day
Started | 68 | 20
Completed | 23 | 8
Not Completed | 45 | 12
Not completed — Lack of Efficacy | 23 | 11
Not completed — Withdrawal by Subject | 6 | 0
Not completed — Other reason | 9 | 1
Not completed — SAE, non-fatal | 1 | 0
Not completed — AE, non-serious non-fatal | 4 | 0
Not completed — SAE, non-fatal+AE, non-serious non-fatal | 1 | 0
Not completed — AE of unknown type | 1 | 0

BASELINE CHARACTERISTICS:
Population: Demographics refer to the Randomized Set (RS).
Arm/Group | Brivaracetam 50 mg/Day | Brivaracetam 100 mg/Day | Total Title
Number analyzed (Participants) | 68 | 20 | 88
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.7 (11.7) | 43.6 (13.2) | 39.0 (12.2)
Age, Customized [Number; unit: participants]
  < 65 years | 66 | 19 | 85
  >= 65 years | 2 | 1 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 8 | 41
  Male | 35 | 12 | 47

OUTCOME MEASURES:

1. Primary Outcome: The Cumulative Exit Rate at 112 Days After the Beginning of the Baseline Antiepileptic Drug (AED) Tapering Phase
Description: The cumulative exit rate was estimated using Kaplan-Meier methods and was based on the duration between start of the Evaluation Period (EP) and the earliest date the first exit criterion was met for each subject. Subjects completing the EP without meeting an exit criterion were censored on Day 112. The primary comparison was BRV 50 mg/day vs a historical control. The upper limit of the 2-sided 95 % Confidence Interval for the estimate was compared to the historical lower bound estimate of 0.722.
Time Frame: From Week 1 up to Week 17
Population: The Efficacy Analysis Set (EFF) consists of all randomized subjects with at least one intake of study medication who also entered into the Baseline antiepileptic drug (AED) Tapering Period and started the withdrawal of Baseline AEDs.
Measure: Number (95% Confidence Interval); unit: proportion of subjects
Groups:
- Efficacy Analysis Set (BRV 50 mg/Day Treated Subjects): The Efficacy Analysis Set (EFF) consists of all randomized subjects with at least one intake of study medication who also entered into the Baseline antiepileptic drug (AED) Tapering Period and started the withdrawal of Baseline AEDs.
Arm/Group | Efficacy Analysis Set (BRV 50 mg/Day Treated Subjects)
Number analyzed (Participants) | 67
proportion of subjects | 0.487 [0.347 to 0.626]

2. Secondary Outcome: The Number of Patients Reporting at Least One Treatment-Emergent Adverse Event (TEAE) During the Course of the Study
Time Frame: Baseline through Re-conversion (approximately 31 weeks)
Population: The Intention-to-Treat (ITT) Set consists of all randomized subjects with at least one intake of study medication.
Measure: Number; unit: Participants
Arm/Group | Brivaracetam 50 mg/Day | Brivaracetam 100 mg/Day
Number analyzed (Participants) | 68 | 20
Participants | 53 | 11

3. Secondary Outcome: The Number of Patient Withdrawal Due to Adverse Events (AEs) During the Course of the Study
Time Frame: Baseline through Re-conversion (approximately 31 weeks)
Population: The Intention-to-Treat (ITT) Set consists of all randomized subjects with at least one intake of study medication.
Measure: Number; unit: Participants
Arm/Group | Brivaracetam 50 mg/Day | Brivaracetam 100 mg/Day
Number analyzed (Participants) | 68 | 20
Participants | 9 | 2

4. Secondary Outcome: The Number of Patients Reporting at Least One Serious Adverse Event (SAE) During the Course of the Study
Time Frame: Baseline through Re-conversion (approximately 31 weeks)
Population: The Intention-to-Treat (ITT) Set consists of all randomized subjects with at least one intake of study medication.
Measure: Number; unit: Participants
Arm/Group | Brivaracetam 50 mg/Day | Brivaracetam 100 mg/Day
Number analyzed (Participants) | 68 | 20
Participants | 5 | 0

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) were collected from Visit 1 (Week -8) over the BRV Add-On Period and Evaluation Period up to the end of the Re-conversion Follow-up Period (Week 23).
Description: Adverse Events refer to the Intention-to-Treat (ITT) Set consisting of all randomized subjects with at least one intake of study medication.
Arm/Group | Brivaracetam 50 mg/Day | Brivaracetam 100 mg/Day
Serious Adverse Events (participants affected / at risk) | 5/68 | 0/20
Other Adverse Events (participants affected / at risk) | 33/68 | 10/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Brivaracetam 50 mg/Day (N=68) | Brivaracetam 100 mg/Day (N=20)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Grand mal convulsion (Nervous system disorders) | 2 (2) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Loss of consciousness (Nervous system disorders) | 1 (1) | 0 (0)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Status epilepticus (Nervous system disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Brivaracetam 50 mg/Day (N=68) | Brivaracetam 100 mg/Day (N=20)
Nausea (Gastrointestinal disorders) | 3 (3) | 2 (3)
Fatigue (General disorders) | 5 (5) | 2 (2)
Nasopharyngitis (Infections and infestations) | 4 (5) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 6 (7) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
Headache (Nervous system disorders) | 9 (10) | 0 (0)
Convulsion (Nervous system disorders) | 3 (3) | 4 (5)
Somnolence (Nervous system disorders) | 4 (4) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 2 (2)
Anxiety (Psychiatric disorders) | 6 (6) | 1 (1)
Depression (Psychiatric disorders) | 7 (7) | 0 (0)
Insomnia (Psychiatric disorders) | 5 (6) | 0 (0)
Hot flush (Vascular disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days